CLINICAL TRIAL: NCT01687205
Title: Phase 1 Evaluation of the Impact of Coitus on Pharmacokinetics and Pharmacodynamics of Tenofovir 1% Gel Following Pericoital or Daily Gel Dosing
Brief Title: Coital Pharmacokinetics/Pharmacodynamics (PK/PD) of Tenofovir Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Mental Health (NIMH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MTN-011; 3UM1AI068633 (NIH); UM1AI068615 (NIH); 11825 (Other: DAIDS protocol #)
Record Dates: First submitted 2012-08-27; First posted 2012-09-18 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Pharmacokinetics of 1% Tenofovir Gel Following Coitus; Pharmacodynamics of 1% Tenofovir Gel Following Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Single Dose/1 hour before and 1 hour after sex (BAT) Cohort
  Interventions: Drug: 1% Tenofovir Gel
- Group 2 (Active Comparator): Multiple Dose Cohort
  Interventions: Drug: 1% Tenofovir Gel

INTERVENTIONS:
Drug: 1% Tenofovir Gel

SUMMARY:
Study Objectives:

* To assess the impact of coitus (and semen) on the pharmacokinetics of tenofovir 1% gel in female genital tract secretions, vaginal and cervical tissue and rectal tract secretions
* To assess the impact of coitus (and semen) on pharmacodynamics of luminal drug by measuring the anti-HIV-1 activity in CVL samples

Study Summary:

MTN-011 will enroll heterosexual monogamous, sexually active couples, in which both partners are healthy and HIV-negative. The female participants must be between the ages of 21-46 (inclusive) and currently using effective non-barrier contraception. Male participants must be 21 years of age or older. This Phase 1 expanded safety study will assess tenofovir PK in the genital tract secretions (CVL), rectal (rectal sponge) and both intracellular and extracellular tissue compartments (vaginal biopsy) in the absence of, or following coitus. Pharmacodynamics (antiviral activity) will also be assessed in CVL. MTN-011 will study the timing in which coitus might have the greatest impact on these variables, which is when gel is applied shortly prior to coitus in the absence of a drug reservoir.

MTN-011 will examine PK/PD in response to a single dose of 1% tenofovir gel applied shortly before sex and compare to PK/PD assessments following a single gel application without sex. Additionally, data obtained from a visit in which participants do not dose with gel and do not have sex will serve as an additional control for the pharmacodynamic (PD) studies of the antiviral activity in CVL. If tenofovir retains its antiviral activity following sex, then the anti-HIV activity in CVL collected at the visit in which female participants dose with gel and have sex should be comparable to that of CVL collected at the visit in which females dose with gel and then do not engage in intercourse and significantly greater than the endogenous anti-HIV activity in CVL obtained at the visit in which participants do not dose with gel but do have sex and the visit in which no gel is administered and sex does occur. Data analysis performed after the completion of enrollment and follow-up procedures will demonstrate if there is an impact of coitus and semen on PK/PD when a single 1% tenofovir dose is applied shortly prior to sex.

ELIGIBILITY:
Inclusion Criteria:

Men and women must meet the following criteria to be eligible for inclusion in the study:

1. Able and willing to provide the following:

   * Written informed consent to be screened for and take part in the study
   * Adequate locator information, as defined in site SOPs
2. Per participant report, at low risk for HIV/STI. Low risk is defined as:

   * No sexually transmitted infections (STIs) in the 6 months prior to Screening
   * No non-therapeutic intravenous drug use in the 18 months prior to Screening
   * In a mutually monogamous relationship with a partner of the opposite sex for 6 months prior to Screening and the intent to stay in this relationship for the next 4 months
3. At Screening and Enrollment, both partners independently report not using barrier contraception and/or barrier protection as part of normal coital routine and report the intent to continue said sexual practice for the duration of study participation
4. HIV-uninfected based upon testing performed by study staff at Screening (per protocol algorithm)
5. Agrees not to participate in other research studies involving drugs, medical devices, or genital and rectal products, or large blood draw studies during study participation
6. Women must also meet the following criteria:

   * Age 21 through 46 years (inclusive) at Screening, verified per site SOPs
   * Pap result in the 12 calendar months prior to Screening consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009), or satisfactory evaluation with no treatment required of non-Grade 0 Pap result per American Society for Colposcopy and Cervical Pathology (ASCCP) guidelines in the 12 calendar months prior to the Screening Visit

   Note: Women with a documented normal result within the 12 months prior to screening need not have a Pap smear during the screening period. Women with abnormal Pap smears can be enrolled upon completion of the initial phase of evaluation if no current treatment is indicated (based on local standard of care for management of abnormal cervical cytology). Need for a repeat Pap within 6 months does not preclude enrollment prior to that result becoming available.
   * Must be currently using effective non-barrier contraception, other than a contraceptive vaginal ring, for at least three months prior to Screening (i.e., oral contraceptive, patch, injectable hormones, subdermal implants, intrauterine device, female or male sterilization) and intending to use this method for the course of the study
   * Per participant report, regular menstrual cycles with at least 21 days between menses (does not apply to participants who report using a progestin-only method of contraception at screening, e.g., Depo-Provera)

   Note: This criterion is not applicable to participants using continuous combination oral contraceptive pills, as the absence of regular menstrual cycles is an expected, normal consequence in this context.
   * Anatomy sufficient for performing pelvic examinations and for collecting vaginal and cervical specimens
   * Female participants must also agree to abstain from intercourse (oral, anal, or penile-vaginal) and other vaginal practices (e.g., masturbation, douching, tampon use, application of lubricants/spermicides or other related practices) 72 hours prior to each follow-up visit.
7. Men must also meet the following criteria:

   * Age 21 or older at Screening, verified per site SOPs
   * Agree to abstain from intercourse (oral, anal, or penile-vaginal) and other penile practices (e.g., masturbation, application of lubricants/spermicides or other related practices) 72 hours prior to each follow-up visit.

Exclusion Criteria:

Men and women who meet any of the following criteria will be excluded from the study.

1. Participant report of any of the following:

   * Known allergy to the study product (ever)
   * Post-exposure prophylaxis (PEP) for HIV exposure within 6 months prior to Screening
   * Participation in any other research study involving drugs, medical devices, or genital products 30 days or less prior to Enrollment
   * Plans to relocate away from the study site in the next 4 months
   * History of domestic violence with current partner (ever)
   * Systemic or topical antimicrobials within the last 7 days prior to Enrollment
   * Currently using or planning to use pharmacologic immune modulator(s)
2. At Screening or Enrollment, symptomatic urinary tract infection (UTI)

   Note: Otherwise eligible participants diagnosed with UTI during screening are offered treatment and may be enrolled after completing treatment and all symptoms have resolved as long as treatment is completed and all symptoms have resolved within 30 days of obtaining informed consent for Screening/Enrollment.
3. At Screening, has a positive hepatitis B surface antigen (HBsAg) test result
4. At Screening or Enrollment, has an STI or reproductive tract infection (RTI) requiring treatment per current Centers for Disease Control (CDC) guidelines
5. Genital signs and/or symptoms of Grade 2 or higher

   Note: For female participants, cervical bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the IoR/designee is considered expected non-menstrual bleeding and is not exclusionary.

   Note: Otherwise eligible participants with exclusionary genital findings may be enrolled after the findings have improved to a non-exclusionary severity grading or resolved as long as treatment is completed and all symptoms have resolved within 30 days of obtaining informed consent for Screening/Enrollment.
6. Has any other condition that, in the opinion of the Investigator of Record (IoR)/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives
7. Women who meet any of the following criteria will be excluded from the study:

   * Participant report (or clinical finding) of the following:

     * Last pregnancy outcome 90 days or less prior to Enrollment
     * Currently pregnant

   Note: Self-reported pregnancy is adequate for exclusion from the study. A documented negative pregnancy test performed by study staff is required for inclusion.
   * Currently breastfeeding
   * Intends to become pregnant in the next 4 months
   * Gynecologic or genital procedure (e.g., tubal ligation, dilation and curettage) within the prior 30 days to Enrollment

   Note: This does not include biopsy for the evaluation of an abnormal pap result or endometrial biopsy that occurred more than 7 days prior to Enrollment.
   * Any of the following laboratory abnormalities at Screening:

     * Hemoglobin less than 10.0 g/dl
     * Platelet count less than 100,000/mm3

   Note: Otherwise eligible participants with an exclusionary test may be re-tested during the screening process
   * Use of a vaginal douche or other intravaginal products (excluding tampon use) in the 30 days prior to Enrollment
   * Currently menopausal or perimenopausal
8. Men who meet any of the following criteria will be excluded from the study:

   * Participant report of penile procedures (e.g. biopsy, circumcision) within 42 days prior to Enrollment
   * For uncircumcised men, per participant report, treatment of candidal balanoposthitis/ balanitis within 30 days prior to Enrollment

Ages: 21 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of tenofovir 1% gel | Visits 3b, 4b, 5b, 6b and 7b.
  To assess the impact of coitus (and semen) on the pharmacokinetics of tenofovir 1% gel in female genital tract secretions, vaginal and cervical tissue and rectal tract secretions
Pharmacodynamics of luminal drug | Visits 2b, 3b, 4b, 5b, 6b and 7b.
  To assess the impact of coitus (and semen) on pharmacodynamics of luminal drug by measuring the anti-HIV-1 activity in CVL samples

SECONDARY OUTCOMES:
Acceptability | Visit 7b.
  To assess the acceptability of the MTN-011 trial to male and female participants

OTHER OUTCOMES:
Impact of coitus and/or tenofovir on the genital tract mucosal environment | Visits 1, 2b, 3b, 4b, 5b, 6b and 7b.
  To assess the impact of coitus and/or tenofovir on the genital tract musical environment
Semen biomarker | Visits 1, 2b, 3b, 5b and 7b.
  To determine whether a semen biomarker can be used to estimate the volume of ejaculate within CVL
Retained drug levels in the lumen | Visits 1, 2b, 3b, 4b, 5b, 6b and 7b.
  To assess whether sufficient drug is retained in the lumen in the absence of or following coitus to inhibit HSV-2 as an additional surrogate biomarker of pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Herold, MD, Study Chair — Albert Einstein College of Medicine; Beatrice A. Chen, MD, MPH, Principal Investigator — University of Pittsburgh; Robert A. Salata, MD, Principal Investigator — Case Western Reserve University
Locations (2):
- United States (2):
  - Case Western Reserve University, Cleveland, Ohio
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Herold BC, Chen BA, Salata RA, Marzinke MA, Kelly CW, Dezzutti CS, McGowan I, Galaska B, Levy L, Piper JM, Hillier S, Hendrix CW. Impact of Sex on the Pharmacokinetics and Pharmacodynamics of 1% Tenofovir Gel. Clin Infect Dis. 2016 Feb 1;62(3):375-382. doi: 10.1093/cid/civ913. Epub 2015 Oct 27. PMID 26508513